CLINICAL TRIAL: NCT05474313
Title: PrEP-3D RCT: A Randomized Controlled Trial Evaluating An Integrated Pharmacy Digital Diary and Delivery Strategy to Increase PrEP Use Among Persons Assigned Male at Birth Who Have Sex With Persons Assigned Male at Birth
Brief Title: A Study Evaluating An Integrated Pharmacy Digital Diary and Delivery Strategy to Increase PrEP Use Among MSM and TGW
Acronym: PrEP-3D RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: San Francisco Department of Public Health (Other Government); Alto Pharmacy (Unknown)
Responsible Party: Principal Investigator, Susan Buchbinder, Director, Bridge HIV, SFDPH, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-35533
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: HIV Prevention; Pre-exposure Prophylaxis (PrEP); Risk Reduction; Adherence, Medication
Keywords: PrEP; pre-exposure prophylaxis (PrEP); Adherence; HIV Risk Reduction; Mobile App; Pharmacy
MeSH Terms: conditions — Risk Reduction Behavior; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrEP-3D (Experimental): Use of Alto Pharmacy, PrEP-3D mobile app and home laboratory testing.
  Interventions: Behavioral: PrEP-3D package
- Control Arm (Other): Participants in the control arm will receive standard of care PREP navigation.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: PrEP-3D package — A package of support tools for accessing, adhering to, and monitoring PrEP use, including Alto Pharmacy delivery services, PrEP-3D mobile app, and home laboratory testing.
  Arms: PrEP-3D
Behavioral: Standard of Care — Participants are given local standard of care navigation for initiation of PrEP
  Arms: Control Arm

SUMMARY:
The PrEP 3D randomized controlled trial (RCT) will study the effectiveness of the PrEP-3D app compared to standard of care for starting pre-exposure prophylaxis (PrEP), continuing PrEP, and adherence to PrEP.

DETAILED DESCRIPTION:
The investigators will be testing a pharmacist-led model of PrEP delivery combined with mobile app-based PrEP support developed by the investigator's team to improve PrEP initiation and persistence. Alto Pharmacy is a full-service online pharmacy already using mobile and web apps to communicate with patients, providers, laboratories, and insurers to provide timely medication delivery. Alto can provide PrEP prescriptions, order laboratory tests, and perform clinical referrals through a collaborative practice agreement (CPA) with SFDPH that allows transfer of these responsibilities. The investigators have integrated online tools with Alto Pharmacy's technology platform to create PrEP-3D: Digital Diary and Delivery, combining a tailored online support tool with the personalized service of a community pharmacy and the convenience of medication delivery. By removing the requirement for initiation and quarterly visits with a primary care physician for PrEP, the PrEP-3D model will expand access to PrEP visits (including for persons who choose not to go to their primary care provider for PrEP) and reduce burden on the health care system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Assigned male at birth who reports sex with persons assigned male at birth
* Willing and able to provide written informed consent
* HIV-uninfected by negative 4th generation HIV test during screening
* Owns a smartphone and has private access to the internet
* Able to understand, read, and speak English or Spanish
* Lives in California
* Self-reported evidence of being at-risk for HIV acquisition, including at least one of the following in the past 6 months:

  * ≥ 1 episode of anal/vaginal sex with a male or transgender female partner;
  * Diagnosed with a bacterial sexually transmitted infection (STI).
* Interested in taking daily TDF/FTC or TAF/FTC PrEP
* Willing and able to receive PrEP prescriptions through Alto Pharmacy (e.g., no specific pharmacy required by health plan, such as Kaiser HMO)
* Creatinine clearance >30 mL/min
* No contraindications to TDF/FTC or TAF/FTC use

Exclusion Criteria:

* Repeatedly reactive HIV test at screening or enrollment
* Signs or symptoms of acute HIV infection at screening or enrollment
* Currently enrolled in another HIV intervention study.
* Unable to commit to study participation for the duration of the study
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of PREP-3D on PREP use | 12 months
  Measurement of PrEP adherence using dried blood spot measurements of tenofovir-diphosphate (TFV-DP) levels greater than or equal to 700 fmol/punch

CONTACTS AND LOCATIONS:
Overall Officials: Susan Buchbinder, MD, Principal Investigator — Bridge HIV, San Francisco Department of Public Health
Locations (2):
- United States (2):
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - Alto Pharmacy, San Francisco, California

IPD SHARING:
Plan to Share IPD: No